CLINICAL TRIAL: NCT06421987
Title: Cardiopulmonary Function and Cerebral Blood Flow in Hodgkin Lymphoma Survivors
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HODNIRS; NCI-2024-03932 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-05-01; First posted 2024-05-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Hodgkin Disease | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SURVIVOR: A survivor of Hodgkin Lymphoma (HL) treated with chest radiation and bleomycin at St. Jude Children's Research Hospital.
  and Control: Voluntarily taking part in this study because you are a relative, friend or employee of St. Jude Children's Research Hospital.
  Interventions: Device: Near Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) — NIRS is a portable, non-invasive, brain imaging device.

SUMMARY:
SURVIVORS

Study participants are being asked to take part in this research study called HODNIRS because the participant is a survivor of Hodgkin Lymphoma (HL) treated with chest radiation and bleomycin at St. Jude Children's Research Hospital. The study is being done to help investigators understand the link between long term effects of chest radiation and bleomycin for HL and brain function in survivors.

Primary Objective To evaluate dynamic changes in CBF and oxygenation during exercise with Near Infrared Spectroscopy (NIRS) in HL survivors and non-cancer controls matched for age, sex, race, and ethnicity. .

Secondary Objectives To examine the degree of CO2 clearance (DLCO/ETCO2) during rest and exercise in Hodgkin Lymphoma (HL) survivors compared to non-cancer controls matched for age, sex, race, and ethnicity.

CONTROLS

Volunteers are being asked to take part in this research study because they are non-first degree relative or friend of someone who received treatment for a childhood cancer or similar illness at St. Jude Children's Research Hospital or are an employee/affiliate of St. Jude Children's Research Hospital and have agreed to be a St. Jude Life Cohort Study (SJLIFE) community control.

DETAILED DESCRIPTION:
NIRS is a portable, non-invasive, brain imaging device that uses low levels of non-ionizing light to record variations in blood flow in the brain. The NIRS is wearable and can read blood flow to the brain during physical activity.

ELIGIBILITY:
Inclusion Criteria:

HL Survivors

* Completed bleomycin and/or thoracic radiation therapy for HL at SJCRH.
* <21-years old at diagnosis; currently ≥18-years of age and ≥2-years post therapy.
* SJLIFE or ACT/SJLIFE participants
* English language proficiency.

Community Controls

* SJLIFE control.
* ≥18-years of age at the time of enrollment with age sampling to broadly match the HL survivors.

Exclusion Criteria:

HL Survivors

* History of cranial or total-body irradiation therapy.
* History of intrathecal or high dose intravenous antimetabolite therapy.
* History of head injury or diagnosis of a genetic disorder associated with cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Near-Infrared Spectroscopy (NIRS) | Baseline
  a non-invasive imaging technology that is used to measure regional or global cerebral tissue oxygenation and cerebral blood flow (CBF) during exercise. NIRS takes advantage of the fact that oxygenated blood and de-oxygenated blood absorb light differently. By measuring the reflected light from blood, the concentration of both oxygenated hemoglobin (HbO2) and deoxygenated hemoglobin (HbdO2) using the modified Beer-Lambert Law can be calculated.

SECONDARY OUTCOMES:
Cardiopulmonary Exercise Testing (CPX) | Baseline
  Cardiopulmonary Exercise Testing (CPX) will be performed with the goal of maximal exertion. Participants are monitored with 12-lead electrocardiogram (ECG) and serial blood pressure measurements during and after exercise, and during recovery. Study participants whose physical performance does not permit walking safely on the treadmill, will perform CPX on a bicycle or upper extremity ergometer using a comparable testing protocol.
  Oxygen consumption during CPX- Oxygen will be measured at baseline and continuously during CPX. Total minute ventilation (respiratory rate X tidal volume; l/min), and ventilatory reserve (l/min) will be used to assess the ability of the pulmonary system to respond to exercise.
Pulmonary Function Testing | Baseline
  As part of the St. Jude Life (SJLIFE) study visit, participants will complete PFT's performed in a single laboratory according to the American Thoracic Society Task Force Guidelines. Pulmonary Function Tests (PFTs) will include:
  1. Forced vital capacity (FVC) - measured in liters
  2. Forced expiratory volume in 1 second (FEV1) - measured in liters/per second
  3. FEV1/FVC ratio - measurement will be a percent.
  4. DLCO capacity of lung to transfer carbon monoxide - measured in mL/min/mm Hg.
  These measurements will be compared with those predicted for the participant's age, race, sex, and height.
Neurocognitive Outcomes | Baseline
  - As part of the SJLIFE study visit, participants will complete neurocognitive testing (Wechsler Abbreviated Scale of Intelligence; Connors Continuous Performance; California Verbal Learning; Coding Digital Symbol; Grooved Pegboard; Trail Making; Verbal Fluence; Visual Selective; Digital Span; and Rey Complex). All tests are converted to z-scores (1.0 z-score is 1 standard deviation lower than the mean).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Phillips, PhD, Principal Investigator — St. Jude
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols